CLINICAL TRIAL: NCT00076232
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Trial of Acyclovir for the Reduction of HIV Acquisition Among High-Risk HSV-2 Seropositive, HIV Seronegative Individuals
Brief Title: A Study of Acyclovir to Help Prevent HIV Infection in People With Genital Herpes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Rona Siskind, DAIDS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HPTN 039; 1R01AI052054 (NIH); 5U01AI047981-05 (NIH); DAIDS-ES ID 10066; NCT00068965 (obsolete NCT alias)
Record Dates: First submitted 2004-01-15; First posted 2004-01-16 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections; HIV Seronegativity; Herpes Genitalis
Keywords: HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Herpes Genitalis | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants will receive acyclovir for the duration of the study
  Interventions: Drug: Acyclovir
- 2 (Placebo Comparator): Participants will receive acyclovir placebo for the duration of the trial
  Interventions: Drug: Acyclovir placebo

INTERVENTIONS:
Drug: Acyclovir — 400 mg tablet taken orally twice daily
  Arms: 1
Drug: Acyclovir placebo — Oral tablet taken twice daily
  Arms: 2

SUMMARY:
Genital herpes (HSV-2) is the most common cause of genital sores worldwide, and the presence of genital sores is a significant risk factor for becoming infected with HIV. This study will test the effectiveness of twice-daily dosing of acyclovir, a commonly prescribed anti-herpes drug, in preventing HIV infection in HSV-2 infected women who sleep with men (WSM) and men who sleep with men (MSM).

Study hypothesis: Given that genital herpes is a significant risk factor to HIV acquisition, twice-daily HSV-2 suppressive therapy - 400 mg of acyclovir - will prevent HIV infection among high risk, HSV-2 seropositive WSM and MSM.

DETAILED DESCRIPTION:
Many studies have shown that prior HSV-2 infection is associated with an increased risk for HIV infection. Acyclovir is the most widely studied and clinically utilized antiviral for the suppression of HSV-2 infection. This study will evaluate the efficacy of twice-daily dosing of acyclovir in preventing HIV infection in both WSM and MSM with genital herpes. For this study, WSM will be enrolled in Lusaka, Zambia; Harare, Zimbabwe; and Johannesburg, South Africa; MSM will be enrolled in Lima and Pucallpa, Peru; Seattle, Washington, USA; New York City, New York, USA; and San Francisco, California, USA.

Participants will be enrolled for 12 months in this study and will be randomly assigned to one of two study arms. The first arm will receive 400 mg acyclovir twice daily; the second arm will receive placebo. Follow-up visits will occur monthly. Participants will be tested for STDs, including HIV and syphilis, at each visit and treated as necessary; participants will also be given adherence and condom counseling, risk behavior and sexual history questionnaires, and genital symptoms questionnaires at all study visits. Medical history will be assessed and participants will undergo blood work at Months 3, 6, 9, and 12.

ELIGIBILITY:
Inclusion Criteria For All Participants:

* HIV-uninfected
* HSV-2 infected
* Plans to stay in the area for the duration of study participation
* Willing and able to provide consent, undergo clinical evaluations, take study drugs, adhere to follow-up schedule, and provide adequate locator information

Inclusion Criteria for MSM:

* At least 1 episode of anal intercourse with another man within 6 months of study entry

Inclusion Criteria for WSM:

* At least 1 episode of unprotected vaginal sex within 6 months of study entry

Exclusion Criteria For All Participants:

* Current enrollment in another HIV vaccine or prevention trial
* History of adverse reaction to acyclovir
* Current or planned use of famiciclovir, valacyclovir, or acyclovir for genital HSV. Use of short-course antiviral therapy for herpes zoster after enrollment is allowed.
* Known plans for travel away from study site for more than 2 months

Exclusion Criteria for MSM:

* In a mutually monogamous relationship with an HIV uninfected partner throughout the past 2 years
* Reported sex at birth as female

Exclusion Criteria for WSM:

* Pregnancy at screening or enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3682 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Serologically confirmed HIV infection | Throughout study

SECONDARY OUTCOMES:
Occurrence and frequency of genital ulcers | Throughout study
Proportion of doses missed by study participants assigned to twice-daily acyclovir and twice-daily placebo | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Study Chair — University of Washington; Anna Wald, MD, MPH, Study Chair — University of Washington
Locations (3):
- United States (3):
  - San Francisco Department of Public Health, AIDS Office, Research Section, San Francisco, California
  - New York Blood Center, New York, New York
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Bruisten SM. Genital ulcers in women. Curr Womens Health Rep. 2003 Aug;3(4):288-98. PMID 12844451
- [Background] Mbopi-Keou FX, Robinson NJ, Mayaud P, Belec L, Brown DW. Herpes simplex virus type 2 and heterosexual spread of human immunodeficiency virus infection in developing countries: hypotheses and research priorities. Clin Microbiol Infect. 2003 Mar;9(3):161-71. doi: 10.1046/j.1469-0691.2003.00550.x. PMID 12667248
- [Background] Schacker T. The role of HSV in the transmission and progression of HIV. Herpes. 2001 Jul;8(2):46-9. PMID 11867018
- [Background] Wald A, Link K. Risk of human immunodeficiency virus infection in herpes simplex virus type 2-seropositive persons: a meta-analysis. J Infect Dis. 2002 Jan 1;185(1):45-52. doi: 10.1086/338231. Epub 2001 Dec 14. PMID 11756980
- [Result] Celum C, Wald A, Hughes J, Sanchez J, Reid S, Delany-Moretlwe S, Cowan F, Casapia M, Ortiz A, Fuchs J, Buchbinder S, Koblin B, Zwerski S, Rose S, Wang J, Corey L; HPTN 039 Protocol Team. Effect of aciclovir on HIV-1 acquisition in herpes simplex virus 2 seropositive women and men who have sex with men: a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Jun 21;371(9630):2109-19. doi: 10.1016/S0140-6736(08)60920-4. PMID 18572080
- [Result] Reid SE, Dai JY, Wang J, Sichalwe BN, Akpomiemie G, Cowan FM, Delany-Moretlwe S, Baeten JM, Hughes JP, Wald A, Celum C. Pregnancy, contraceptive use, and HIV acquisition in HPTN 039: relevance for HIV prevention trials among African women. J Acquir Immune Defic Syndr. 2010 Apr;53(5):606-13. doi: 10.1097/QAI.0b013e3181bc4869. PMID 19838129
- [Result] Watson-Jones D, Wald A, Celum C, Lingappa J, Weiss HA, Changalucha J, Baisley K, Tanton C, Hayes RJ, Marshak JO, Gladden RG, Koelle DM. Use of acyclovir for suppression of human immunodeficiency virus infection is not associated with genotypic evidence of herpes simplex virus type 2 resistance to acyclovir: analysis of specimens from three phase III trials. J Clin Microbiol. 2010 Oct;48(10):3496-503. doi: 10.1128/JCM.01263-10. Epub 2010 Aug 11. PMID 20702659
- [Result] Curlin ME, Cassis-Ghavami F, Magaret AS, Spies GA, Duerr A, Celum CL, Sanchez JL, Margolick JB, Detels R, McElrath MJ, Corey L. Serological immunity to adenovirus serotype 5 is not associated with risk of HIV infection: a case-control study. AIDS. 2011 Jan 14;25(2):153-8. doi: 10.1097/QAD.0b013e328342115c. PMID 21150554
- [Result] Jacob ST, Baeten JM, Hughes JP, Peinado J, Wang J, Sanchez J, Reid SE, Delany-Moretlwe S, Cowan F, Fuchs JD, Koblin B, Griffith S, Wald A, Celum C. A post-trial assessment of factors influencing study drug adherence in a randomized biomedical HIV-1 prevention trial. AIDS Behav. 2011 Jul;15(5):897-904. doi: 10.1007/s10461-010-9853-2. PMID 21104007
- [Result] Sanchez J, Sal Y Rosas VG, Hughes JP, Baeten JM, Fuchs J, Buchbinder SP, Koblin BA, Casapia M, Ortiz A, Celum C. Male circumcision and risk of HIV acquisition among MSM. AIDS. 2011 Feb 20;25(4):519-23. doi: 10.1097/QAD.0b013e328340fd81. PMID 21099672
- [Derived] Fuchs J, Celum C, Wang J, Hughes J, Sanchez J, Cowan F, Reid S, Delany-Moretlwe S, Corey L, Wald A; HIV Prevention Trials Network 039 Protocol Team. Clinical and virologic efficacy of herpes simplex virus type 2 suppression by acyclovir in a multicontinent clinical trial. J Infect Dis. 2010 Apr 15;201(8):1164-8. doi: 10.1086/651381. PMID 20214474